CLINICAL TRIAL: NCT00501683
Title: A Mass Balance Study to Investigate the Metabolic Disposition of a 400 mg Single, Oral Dose of GSK189075 in Healthy Male Subjects
Brief Title: A Single Dose Of GSK189075 Taken By Mouth Containing Small Amounts Of Radioactivity Studied In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KG2105264
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: metabolite profiling; excretion,; radioactivity,; pharmacokinetic,; mass balance,
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Radiolabelled GSK189075

SUMMARY:
This study will look at the relative amounts of GSK189075 that are found in samples of blood, urine, and feces of healthy male volunteers. Results of the study will be used to understand how the drug is converted in the body and how it is eliminated.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy, non-smoking male.
* Are 30 to 55 years old, inclusive.
* Have a Body Mass Index (BMI) between 19-30 kg/m2, inclusive; and a body weight >110 lbs.
* Have a history of regular bowel movements (at least 4 times per week).
* Are willing and able to provide written informed consent before the start of any study-related procedures.

Exclusion Criteria:

* Have any significant laboratory abnormality or history of liver or kidney disease.
* Have any significant abnormality in your electrocardiograms (ECG) which are recordings of your heart rhythm.
* Have a current condition(s) that alters normal gastrointestinal (GI) function (such as constipation or removal of your gallbladder).
* Have an illness that requires treatment by a physician in the 30 days before screening or a fever and illness in the 5 days before dosing.
* Have blood pressure that is outside the normal range.
* Have a resting pulse rate that is outside the normal range.
* Have had surgery within 3 months before screening, unless approved by the GSK medical monitor.
* Have a drug allergy which the investigator feels would make it unsafe for you to participate in the study.
* Have a history of or current abuse of alcohol.
* Have a history of or current use of illicit drugs, or a positive drug screen.
* Have used tobacco products within 3 months prior to screening or have a positive cotinine test result.
* Are unable to refrain from foods or beverages containing coffee, tea, or chocolate for 72 hours before dosing with study drug and until 24 hours after dose.
* Have a positive test for human immunodeficiency virus (HIV) antibody or hepatitis B surface antigen or hepatitis C antibody.
* Have taken prescription or non-prescription drugs, including vitamins, herbal products, or plant-derived supplements (including St John's Wort) within 14 days (or less than 5 half-lives) before the first dose of study medication, unless approved by the GSK medical monitor
* Have participated in an investigational drug study within the 30 days before screening, or participated within the last 12 months in a study with another radio labeled drug product.
* Have a total radiation exposure from the previous 3-year period that is over 10 mSv (either from your work or through participation in other research studies). Clinical (therapeutic or diagnostic) exposure will not be included.
* Have donated blood (450 mL or more) within the previous 12 weeks.
* Are in an occupation which requires monitoring for radiation exposure, nuclear medicine procedures or have had excessive x-rays within the past 12 months.
* Are not able to follow the study directions.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2006-11

PRIMARY OUTCOMES:
Laboratory tests to determine the amount of radiolabelled drug that is found in blood, urine, and feces. Blood samples at Days 1-5. | at Days 1-5.
Urine & Fecal collection at Day -1 & days 1-5. | at Day -1 & days 1-5.

SECONDARY OUTCOMES:
Adverse events (AEs), vital signs, ECGs and clinical laboratory assessments at each day for up to 10 days | at each day for up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States